CLINICAL TRIAL: NCT01647711
Title: A Phase 1b Study of Intermittent Administration of High Doses of the Irreversible EGFR Inhibitor Afatinib as a Means of Achieving Plasma Levels Active Against Non-small Cell Lung Cancer With Known T790M Mutations
Brief Title: A Study of Intermittent, High-dose Afatinib to Determine the Maximal Tolerated Dose and Assess Activity of This Dose Against Non-small Cell Lung Cancer With T790M Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.121
Record Dates: First submitted 2012-07-16; First posted 2012-07-23 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Maximum Tolerated Dose

ARMS (1):
- Afatinib (Experimental): Establish the Maximal Tolerated Dose of a pulsatile, high-dose regimen of afatinib in patients with advanced solid tumors followed by treatment at that dose or a lower dose in patients with stage IV non-small cell lung cancer harboring EGFR T790M mutations who have progressed on therapy with a reversible tyrosine kinase inhibitor
  Interventions: Drug: Dose escalation followed by treatment with MTD

INTERVENTIONS:
Drug: Dose escalation followed by treatment with MTD — Fixed 3+3 dose escalation; expansion of MTD cohort

SUMMARY:
This trial is divided into Part A and Part B. The primary objective of Part A is to establish the Maximal Tolerated Dose of intermittent high dose afatinib. The primary objective of Part B is to assess the response rate of patients with non-small cell lung cancer with EGFR T790M mutations to a dose of intermittent afatinib established in Part A.

The secondary objective is to explore tumor response and tumor-derived biological markers of response to afatinib, as well as pharmacokinetic parameters of afatinib.

ELIGIBILITY:
Inclusion criteria:

Part A only:

1. Patients with histologically confirmed advanced solid tumours that are metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Patients who refuse standard therapy are also eligible.

   Part B only:
2. Pathologically confirmed diagnosis of Stage IV (M1a or b) non-small cell lung cancer
3. Documented Epidermal Growth Factor Receptor (EGFR) T790M mutation
4. Progression of disease on a reversible tyrosine kinase inhibitor within 30 days of starting study drug. Loss of exposure to prior EGFR TKI should not be >30 days; any procedural delay in confirmation of progression is to be discussed with the BI Clinical Monitor.

   Parts A and B:
5. Evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Age >/= to 18 years
7. Eastern Cooperative Group (ECOG) performance status 0-1
8. Adequate organ function
9. Recovered from any previous therapy-related toxicity to </= to Grade 1 at study entry (except for stable sensory neuropathy </= Grade 2 and alopecia)
10. Written informed consent
11. Ability to take oral medication

Exclusion criteria:

Parts A and B:

1. Chemotherapy, biological therapy, or investigational agents (except erlotinib or gefitinib) within 4 weeks prior to the start of study treatment
2. Hormonal treatment within 2 weeks prior to the start of study treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer is permitted)
3. Radiotherapy within two weeks prior to the start of study treatment (except palliative radiotherapy given for symptom control)
4. Less than 3 days from prior treatment with gefitinib or erlotinib. Patients with adverse events related to gefitinib or erlotinib must recover to Grade 1 or less to be eligible.
5. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
6. Known hypersensitivity to afatinib or the excipients of any of the trial drugs
7. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to starting study treatment
8. Women of childbearing potential and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 2 months after treatment has ended.
9. Female patients of childbearing potential who are nursing; are pregnant; are not using an acceptable method of birth control, or do not plan to continue using this method throughout the study; and do not agree to submit to pregnancy testing required by this protocol
10. Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
11. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured
12. Required treatment with any of the prohibited medications listed in this protocol that cannot be stopped for the duration of trial participation
13. Known pre-existing Interstitial Lung Disease
14. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (for example, Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption) in the opinion of the investigator
15. Active hepatitis B infection (defined as the presence of Hepatitis B DNA), active hepatitis C infection (defined as the presence of Hepatitis C RNA) and/or known Human Immunodeficiency Virus carrier
16. Prior participation in a blinded afatinib clinical study, unless permission to unblind was granted in consultation with the Clinical Monitor of the blinded study
17. Meningeal carcinomatosis
18. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued use of corticosteroids or have been on stable doses of corticosteroids for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment
19. QTc interval > 0.47 seconds as measured during screening procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- United States (2):
  - Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - Boehringer Ingelheim Investigational Site, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Afatinib was administered until disease progression, however patients experiencing clinical benefit were allowed to continue treatment for as long as judged beneficial by the investigator.
Groups:
- Afatinib 90mg: Patients received oral administration of afatinib 90mg film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
- Afatinib 120mg: Patients received oral administration of afatinib 120mg film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
- Afatinib 150mg: Patients received oral administration of afatinib 150mg film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
- Afatinib 160mg: Patients received oral administration of afatinib 160mg film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
- Afatinib 200mg: Patients received oral administration of afatinib 200mg film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
Period: Overall Study
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg
Started | 6 | 3 | 9 | 11 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 9 | 11 | 6
Not completed — Progressive disease | 6 | 2 | 6 | 8 | 2
Not completed — Other adverse event | 0 | 0 | 2 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Refused to continue taking medication | 0 | 0 | 0 | 2 | 1
Not completed — Other reason not defined | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who took at least one dose of afatinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg | Total
Number analyzed (Participants) | 6 | 3 | 9 | 11 | 6 | 35
Age, Continuous [Median (Full Range); unit: Years] | 65.0 [64 to 80] | 58.0 [50 to 77] | 65.0 [54 to 77] | 61.0 [45 to 70] | 62.5 [54 to 75] | 64.0 [45 to 80]
Gender [Count of Participants; unit: Participants]
  Female | 2 | 1 | 6 | 10 | 5 | 24
  Male | 4 | 2 | 3 | 1 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities
Description: Percentage of participants with Dose Limiting Toxicities (DLTs), based on investigator assessment, for determination of Maximum Tolerated Dose (MTD). MTD was defined as the dose in which less than 2 of up to 6 patients developed a DLT.
Time Frame: 28 days
Population: Treated set including patients eligible for MTD determination
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 5
Percentage of participants | 16.7 | 0.0 | 0.0 | 0.0 | 40.0

2. Secondary Outcome: Objective Response Rate for Patients With EGFR T790M Mutations
Description: Objective response rate for patients with Epidermal Growth Factor Receptor (EGFR) T790M mutations. Objective response was defined as Complete Response (CR): Disappearance of all target lesion or Partial Response and (PR): >=30% decrease in the sum of the longest diameter of target lesions, according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
  This endpoint was originally planned to be analysed in part B of the study, however as no participants were treated in part B the analysis was performed on the part A participants.
Time Frame: From first drug administration until last drug administration, up to 420 days
Population: Treated set including participants with EGFR T790M positive mutations
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg
Number analyzed (Participants) | 1 | 0 | 7 | 1 | 4
Percentage of participants | 0.0 |  | 14.3 | 0.0 | 0.0

3. Secondary Outcome: Cmax of Afatinib on Day 3 of Course 1
Description: Maximum measured concentration (Cmax) of afatinib as determined on day 3 of course 1 for patients in Part A
Time Frame: 47 hours (h) 55 minutes (min), 49h, 50h, 51h, 52h, 53h, 54h, 55h after first dose administration (on day 3 of course 1)
Population: Pharmacokinetic set which included all patients treated in part A who were documented to have taken at least one dose of afatinib and who had in addition at least one valid afatinib concentration available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg
Number analyzed (Participants) | 6 | 3 | 8 | 8 | 5
ng/mL | 129 (46.2) | 155 (86.9) | 311 (58.8) | 313 (35.6) | 461 (50.3)

4. Secondary Outcome: Determination of Dosage for Expansion Cohort in Part B
Description: Determination of dosage for expansion cohort in Part B. Dosage was the MTD or less depending on tolerability.
Time Frame: 28 days
Population: Treated set including patients eligible for MTD determination
Measure: Number; unit: mg
Groups:
- Afatinib: Patients receiving oral administration of afatinib film-coated tablet once daily for three days, repeated every 14 days, during each 28-day cycle.
Arm/Group | Afatinib
Number analyzed (Participants) | 30
mg | 150

5. Primary Outcome: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD) was defined as the dose in which less than 2 of up to 6 patients developed a Dose Limiting Toxicity (DLT).
Time Frame: 28 days
Population: Treated set including patients eligible for MTD determination
Measure: Number; unit: mg
Arm/Group | Afatinib
Number analyzed (Participants) | 30
mg | 160

ADVERSE EVENTS:
Time Frame: From first treatment administration until 28 days after the last administration, up to 448 days
Groups:
- All Participants: All treated participants included in the study.
Arm/Group | Afatinib 90mg | Afatinib 120mg | Afatinib 150mg | Afatinib 160mg | Afatinib 200mg | All Participants
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 7/9 | 4/11 | 1/6 | 14/35
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 9/9 | 11/11 | 6/6 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 90mg (N=6) | Afatinib 120mg (N=3) | Afatinib 150mg (N=9) | Afatinib 160mg (N=11) | Afatinib 200mg (N=6) | All Participants (N=35)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 90mg (N=6) | Afatinib 120mg (N=3) | Afatinib 150mg (N=9) | Afatinib 160mg (N=11) | Afatinib 200mg (N=6) | All Participants (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 2 | 4
Eyelid margin crusting (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 7 | 11 | 6 | 31
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 5
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 5 | 5 | 4 | 16
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 5 | 4 | 13
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Catheter site ulcer (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 2
Fatigue (General disorders) | 3 | 1 | 5 | 7 | 2 | 18
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 7 | 1 | 9
Oedema peripheral (General disorders) | 1 | 0 | 2 | 1 | 1 | 5
Pyrexia (General disorders) | 2 | 0 | 2 | 0 | 0 | 4
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 3 | 0 | 4
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 3 | 0 | 3 | 2 | 1 | 9
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 4 | 4 | 3 | 12
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 5
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vulval haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 0 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3 | 1 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 4 | 4 | 17
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
One patient was screened in part B of the study, the patient did not meet eligibility requirements and was not treated. The trial completed enrollment in Part A before any additional patients were screened for Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.